CLINICAL TRIAL: NCT06477185
Title: Characterization of Tuberculosis Associated Lung Fibrosis and Respiratory Impairment, and Prevention Using Doxycycline in A Double Blind Randomized Controlled Trial
Brief Title: Characterization of Tuberculosis Associated Lung Fibrosis and Respiratory Impairment, and Prevention Using Doxycycline
Acronym: TALF-TB
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: Makerere University Lung Institute (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Mak-SOMREC-2021-177
Record Dates: First submitted 2023-08-10; First posted 2024-06-27 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Tuberculosis, Pulmonary
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — Doxycycline

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention: Doxycycline (Experimental): Oral doxycycline (100 mg) administered once daily for 12 weeks
  Interventions: Drug: Doxycycline
- Control arm (Placebo Comparator): Oral placebo (matching with doxycycline) will be administered once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxycycline — Doxycycline is a bacteriostatic tetracycline antibiotic with ability to immunomodulate matrix metalloproteinases, enzymes well known to cause lung damage via breakdown lung extracellular matrix.
  Arms: Intervention: Doxycycline
Drug: Placebo — This will be a chemically inert substance, designed to match oral doxycycline capsules but with no chemically active ingredients.
  Arms: Control arm

SUMMARY:
The goal of this clinical trial is to assess the efficacy(effectiveness) of doxycycline, a potent inhibitor of matrix metalloproteinase (lung collagenase) activity in prevention of Tuberculosis associated lung fibrosis and associated lung function decline among patients with drug sensitive advanced TB. The main question[s] it aims to answer are:

* Does doxycycline have a significant anti-fibrosis role when given as adjuvant therapy to TB patients with advanced pulmonary TB in a double blind randomized placebo controlled trial?
* How does long term respiratory function defer between patients who received adjuvant doxycycline aimed at prevention of TB associated lung fibrosis and those who received a placebo in a double blind randomized controlled trial?

Participants will be subjected to the following:

* Experimental arm: Doxycycline 100 mg once daily for 12 weeks administered concurrently with standard of care anti-TBs.
* Comparator arm: Placebo once daily for 12 weeks administered concurrently with standard of care anti-TBs.

DETAILED DESCRIPTION:
This will be a double-blind randomized block stratified clinical trial. Participants will be enrolled if they have advanced drug sensitive TB evidenced by infiltrates/lesions in at least 2 zones on a chest X-ray, among other inclusion criteria.

Participants will receive 100mg of doxycycline or matching placebo once a day for 12 weeks in addition to standard anti TB therapy.

Participants will undergo baseline high resolution CT scans to evaluate lung parenchyma involvement and repeat CT scans at 12 months to score TB associated fibrosis.

Lung function assessment with spirometry will be done at 6 and 12 months after enrolment to assess trends of lung function in the control and intervention study arms.

Profibrotic cytokines (TGFbeta) and Matrix metalloproteinases (1, 3 ,8,9) will be measured at baseline , 3 and 6 months after enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 - 65 years
* Index PTB episode (sputum smear positive or GeneXpert positive with rifampicin susceptibility)
* Baseline CXR showing infiltrates in at least 2 lung zones (≥30% lung involvement) meeting criteria for moderate/advanced PTB
* HIV uninfected
* Subjects willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
* Able to give written informed consent.

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Baseline serum creatinine or liver enzymes >2 times above upper limit of normal
* Taking corticosteroids for ≥14 days or anti-TBs >7days
* Prospects already enrolled in another clinical trial
* Diabetic patients (most diabetics are on metformin or have history of metformin use. Metformin is postulated to have an anti-fibrosis role)
* Patients with malignancy or on anticancer medication
* Situation where a participant is taking a drug/medication known to interact with the trial drug.
* Known allergies to doxycycline or other tetracyclines
* Known autoimmune disease
* Any factor felt to significantly increase risk of adverse event

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-12-04 (Actual); Primary Completion 2026-12-20 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Mean High resolution CT (HRCT) fibrosis scores | 12 months
  Quantified fibrosis scores (e.g. 0 - 25) will be derived from the CT interpretation tool, and recorded for each participant at baseline and 12 months' HRCT images, and compiled per treatment arm.
  Mean scores per study arm (intervention and control) will de determined for both baseline and 12 months' HRCT scans.
Efficacy of doxycycline as an anti-TB associated fibrosis agent | 12 months
  This will be estimated or analyzed using analysis of covariance method. The difference in the mean 'total HRCT fibrosis score' between the intervention and control study arms shall be compared at 12 months adjusting for the total scores measured at baseline. A linear regression model shall be fit on log transformed values of total HRCT scores for each individual.

SECONDARY OUTCOMES:
Lung function assessment | 12 months
  Lung volumes including Forced expiratory volume in 1 second (FEV1), Forced vital capacity(FVC) will be obtained at spirometry for all subjects in both study arms (doxycycline and placebo) and compared with predicted values (standardized values for age, sex, race and smoking status) and results (percentage of predicted) compared across both study groups at 6 and 12 months.
Correlation between the High-Resolution CT fibrosis score and lung function assessment | 12 months
  TB associated fibrosis will be quantified on CT using total scores derived a modified and adapted version of the Bhalla CT interpretation score for HRCTs done at baseline and 12 months. Lung function assessment will be by spirometry and will be derived as percentage predicted values of participants' lung volumes (FEV1, FVC) at 6 and 12 months and age, sex, race and smoking status standardized values. To estimate the correlation between the HRCT fibrosis score and the lung function assessment in each study arm (Doxycycline versus placebo); 3 log linear models shall be fit. These will include:
  * Log linear model of interaction between FEV1 and treatment arm
  * Log linear model of interaction between FVC and treatment arm
  * Log linear model of interaction between FEV1/FVC ratio and treatment arm
comparison of trends of cytokines (matrix metalloproteinases and TGF beta) between intervention and control arm | 6 months
  Serum concentrations of matrix metalloproteinases (MMPs 1, 3, 8, 9) and Transforming growth factor beta 1 (TGFβ1) will be measured in ng/ml at baseline, 3 and 6 months. Means of the MMP concentrations will be calculated and compared between intervention and placebo arm (at baseline, 3 and 6 months) and analyzed using repeated analysis of variance and mixed effect model.

CONTACTS AND LOCATIONS:
Locations (2):
- Uganda (2):
  - Makerere University Lung Institute, Kampala, Kampala
  - Mulago National Referral Hospital, Kampala

IPD SHARING:
Plan to Share IPD: Yes
All individual participants' data collected during the trial will be available for sharing after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After end of trial and publication of results
Access Criteria: To any one who requests